CLINICAL TRIAL: NCT00034580
Title: Olanzapine Versus Active Comparator in the Treatment of Bipolar I Disorder, Manic or Mixed
Brief Title: Olanzapine Versus Active Comparator in the Treatment of Bipolar I Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5528; F1D-US-HGJT
Record Dates: First submitted 2002-04-30; First posted 2002-05-01 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Bipolar Disorder
Keywords: Bipolar I Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Olanzapine; Risperidone

INTERVENTIONS:
Drug: olanzapine
Drug: risperidone

SUMMARY:
This is a research study comparing the safety and efficacy of two active study medications for the treatment of bipolar I disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject, 18-70 years of age
* Female subjects of childbearing potential must be using a medically accepted means of contraception
* Each subject must have a level of understanding sufficient to perform all tests and examinations required by the protocol
* Subjects must be considered reliable

Exclusion:

* Female subjects who are either pregnant or nursing
* Uncorrected hypothyroidism or hyperthyroidism
* Narrow-angle glaucoma
* Subjects who present a serious and immediate risk of endangering him or herself

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326
Dates: Start 2001-08; Study Completion 2002-08

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Berkley, California
  - Los Angeles, California
  - Orange, California
  - San Marcos, California
  - Torrance, California
  - Denver, Colorado
  - Middleton, Connecticut
  - Washington D.C., District of Columbia
  - Winter Park, Florida
  - Boise, Idaho
  - Hoffman Estates, Illinois
  - Natick, Massachusetts
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Clementon, New Jersey
  - Olean, New York
  - Philadelphia, Pennsylvania
  - Madison, Tennessee
  - Houston, Texas
  - Richmond, Virginia
  - Roanoke, Virginia